CLINICAL TRIAL: NCT02686996
Title: The Potential of Carnosine Supplementation in Reducing the Cardiometabolic Risk: a Double-blind, Placebo-controlled Trial
Brief Title: The Potential of Carnosine Supplementation in Reducing the Cardiometabolic Risk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Monash University (Other)
Responsible Party: Principal Investigator, Barbora de Courten, Associate Professor, Monash University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 16061A
Record Dates: First submitted 2016-02-09; First posted 2016-02-22 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Insulin Sensitivity
Keywords: carnosine; Insulin sensitivity; low grade inflammation; Oxidative stress; Advanced glycation; Type 2 diabetes; Cardiovascular disease
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2; Cardiovascular Diseases | interventions — Carnosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Each participant will be given a daily oral dose 2 g of carnosine (2 tablets twice daily) for 14 weeks
  Interventions: Dietary Supplement: carnosine
- Control (Placebo Comparator): Each participant will be given a daily oral dose 2 g of identical placebo tablets ( 2 tablets twice daily) for 14 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: carnosine — Carnosine capsules (2g) twice per day for 14 weeks
  Arms: Intervention
Other: Placebo — Placebo (methylcellulose) capsules for control group identical to intervention capsules and dose
  Arms: Control

SUMMARY:
The aim of this study is to determine whether carnosine supplementation in overweight/obese individuals can improve insulin secretion and/or insulin resistance by decreasing sub clinical inflammation.

The investigators hypothesise that carnosine supplementation will reduce type 2 diabetes and cardiovascular risk factors by lowering chronic low-grade inflammation (CLI), oxidative stress, advanced glycation end products (AGEs), and advanced lipoxidation end products (ALEs).

Aim :To determine the capacity of carnosine supplementation to decrease major risk factors for type 2 diabetes and cardiovascular disease and identify metabolic pathways involved, specifically by:

1. Reducing diabetes risk (insulin sensitivity; secretory function and glucose tolerance)
2. Improving cardiovascular risk factors (lipids; arterial (aortic) stiffness; central blood pressure (cBP); endothelial function).
3. Decreasing the CLI, oxidative stress, AGEs, and ALEs, and increase detoxification of reactive carbonyl species (RCSs).

DETAILED DESCRIPTION:
Cardiovascular risk factors including type 2 diabetes underpin a major threat to the globe and result in a heavy health and financial burden across the healthcare system. Treating type 2 diabetes and cardiovascular disease is expensive and often unsatisfactory. Current medications bring unwanted side effects, and often merely delay rather than prevent type 2 diabetes complications and cardiovascular disease. As a further concern, the micro- and macrovascular complications of type 2 diabetes often start developing before actual diagnosis. Diabetes prevention and treatment through weight loss and exercise programs is a difficult and costly public health measure, leaving the tidal wave of type 2 diabetes to swell even more. An alternative is urgently needed: a low-cost safe approach, easy to implement at population level.

Could carnosine be that alternative? The evidence suggests carnosine has significant metabolic impact and presents such an alternative. A naturally occurring dipeptide, carnosine is already emerging as a human therapy in exercise physiology, heart failure, cataract prevention and treatment, neurology, and psychiatry. A promising further use may derive from its effect on cardiovascular risk factors. Metabolic research, though confined to animal studies, strongly suggests that carnosine supplementation aids the prevention and treatment of obesity, type 2 diabetes, and cardiovascular disease - by virtue of its anti-inflammatory, antioxidative, and anti-glycating effects. The investigators conducted the first pilot data in human and demonstrate relationships among carnosine, obesity, insulin resistance, and dyslipidemia. Put briefly, the pilot weighs strongly in favour of carnosine as a means of reducing cardiovascular risk in humans.

Too good to be true? Apart from its excellent side-effect profile, carnosine is inexpensive and seemingly safe (available as an over-the-counter food additive), making it prima facie ideal for population use. In this setting research is now urgently needed - to test the significant metabolic potential of carnosine to address a major health problem.

The investigators propose a comprehensive double-blind placebo-controlled human trial to investigate the effects of carnosine supplementation on cardiovascular risk factors. If the investigators demonstrate a role in reducing risk factors for type 2 diabetes and cardiovascular disease in overweight and obese non-diabetic humans, the public health implications will be revolutionary, offering the world a genuine low cost, accessible, intervention to curtail the advance of obesity, type 2 diabetes, and cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 or <60 years,
* Weight change < 5 kg in last 12 months
* BMI >25kg/m2 but weight <159kg due to DEXA scan restrictions
* Non-diabetic, no allergy, non-smoker, no high alcohol use
* No current intake of medications including vitamin supplements
* No kidney, cardiovascular, haematological, respiratory, gastrointestinal, endocrine or central nervous system disease, as well as no psychiatric disorders, no active cancer within the last five years; no presence of acute inflammation (by history, physical or laboratory examination)
* Not pregnant or lactating

Exclusion Criteria:

* Age <18 or > 60 years
* Weight change > 5 kg in last 12 months
* Diabetes (diagnosed or oral glucose tolerance test (OGTT), allergy
* Current smoking habit, high alcohol use
* Current intake of medications including vitamin supplements
* Kidney, cardiovascular, haematological, respiratory, gastrointestinal, endocrine or central nervous system disease, as well as psychiatric disorder, active cancer within the last five years; presence of acute inflammation (by history, physical or laboratory examination)
* pregnancy or lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2017-02-13 (Actual); Primary Completion 2020-02-13 (Estimated); Study Completion 2020-06-12 (Estimated)

PRIMARY OUTCOMES:
Change in insulin sensitivity measured by euglycaemic glucose clamp | From baseline to 14 weeks
  The clamp will be used to measure insulin sensitivity. The clamp is initiated by an intravenous bolus injection of insulin (9milliUnit/kg). Insulin is then constantly infused at a rate of 40 milliUnit.m-2.min-1 for 120 min into an arm vein, whilst glucose is variably infused to maintain euglycaemia. Plasma glucose values will be monitored every 5 minutes during the clamp and the variable infusion rate of glucose is adjusted to maintain blood glucose at a constant value of 5mmol/L.

SECONDARY OUTCOMES:
Change in markers of endothelial dysfunction | From baseline to 14 weeks
  This is done using non-invasive peripheral arterial tomography (PAT; endothelium-dependent digital pulse amplitude testing (EndoPAT), Itamar Medical Ltd, Israel), which records continuous plethysmo¬graphic signals of the finger arterial pulse wave. Finger plethysmographic probes are placed on each index finger; and after a 5 min equilib¬ration period, a blood pressure cuff on the non-dominant arm is inflated to 60 mmHg above systolic for 5 min and then deflated to induce reactive hyperaemia. Measurements of post-occlusion changes (reactive hyperaemia PAT: RH-PAT) are continued for 10 min. Results are normalised to the non-occluded arm, compensating for potential systemic changes (RH-PAT ratio).
Change in Acute Insulin Secretory Response - Intravenous Glucose Tolerance Test | From baseline to 14 weeks
  This will be measured in response to 25g intravenous glucose and calculated as the average incremental plasma insulin level from the third to the fifth minute after the glucose bolus.
Change in Resting systolic and diastolic blood pressure | From baseline to 14 weeks
  Resting systolic and diastolic blood pressure and pulse rate will be measured using an automated oscillometric measurement system (Dinamap, USA) after a 30 minute rest.

OTHER OUTCOMES:
Change in Arterial waveform measurement | From baseline to 14 weeks
  This is done with the BP+ device (Uscom Ltd, Australia). This is a device for non-invasive measurement of central blood pressure and augmentation index using an oscillometric method.
Change in Oral Glucose Tolerance Test -OGTT | From baseline to 14 weeks
  After a 10-12 h overnight fast, participants will ingest 75g of glucose over 2 mins. Blood samples will be drawn at 0, 30, 60, 90 and 120 min for plasma glucose and insulin concentrations. We will evaluate the area under the curve.
Change in Measure of Adiposity (DEXA) | From baseline to 14 weeks
  body composition by dual energy x-ray absorptiometry (DEXA), which is a non-invasive assessment of soft tissue composition by region with a precision of 4-5%; central adiposity assessed in duplicate using a constant-tension tape for taking waist, and hip circumference. Bioimpedance measurement will be also collected for validation purposes.
Change in plasma and urinary AGEs | From baseline to 14 weeks
  Measured by liquid chromatography-tandem mass spectrometry and ELISA tests. Circulating receptor for AGEs will be measured by ELISA. Protein modifications and the effect of carnosine supplementation will be determined by proteomic approaches.
Change in plasma and urinary ALEs | From baseline to 14 weeks
  This will be determined by measuring the advanced oxidation protein products and by measuring the cysteinate form of albumin by mass spectrometry. Mercapturic acid adducts with the main reactive carbonyls species will also be quantitatively determined by liquid chromatography electrospray ionization mass spectrometry/mass spectrometry analysis (LC-ESI-MS/MS).
Change in inflammatory markers | From baseline to 14 weeks
  Plasma inflammatory markers (interleukin 1β, 6, 8 and 10, tumour necrosis factor α (TNFα), macrophage migration inhibitory factor, monocyte chemotactic protein-1) will be measured by quantitative sandwich enzyme immunoassays (R & D Systems Inc, USA) (interassay Coefficients of Variation: 7.2%, 10.2%, 5.8%, respectively). Plasma C- reactive protein (hsCRP) via a high sensitivity assay (BN-II nephelometer; Dade Behring Diagnostics, NSW).
Change in Carnosine concentrations in skeletal muscle | From baseline to 14 weeks
  This will be measured in skeletal muscle (soleus and gastrocnemius) non-invasively with proton magnetic resonance spectroscopy (1 H-MRS) on a 3 tesla magnetic resonance imaging (3T MRI) scanner (Siemens Trio, Germany) as developed by our group. The lower leg is fixed in a knee coil and single-voxel point-resolved spectroscopy is used: repetition time (TR) 2.000 ms, echo time (TE) 30 ms, 128 excitations. The integral of the second conserved cysteine to histidine (C2H) peak (at 8 ppm) is quantified relative to the water peak integral. We will also measure muscle carnosine content ex-vivo by high performance liquid chromatography (HPLC) from the biopsy samples of vastus lateralis.
Change in Serum and urine carnosine | From baseline to 14 weeks
  This will be quantitatively analysed with HPLC-ESI-MS systems (triple quadrupole orbitrap mass spectrometry analyser); metabolites of carnosine from covalent detoxification of the reactive carbonyl species (precursors of AGEs and ALEs) will be profiled similarly.
Change in Plasma carnosinase protein content | From baseline to 14 weeks
  This will be measured by ELISA for human carnosinase 1 (CN1) with a monoclonal antibody (clone ATLAS, Abcam plc) and peroxidase substrate .
Change in Other Tissue Analyses | From baseline to 14 weeks
  We will measure changes in the expression and activation of important insulin signalling proteins, including the insulin receptor,and we will measure inflammation markers in skeletal, muscle and adipose tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Barbora de courten, MD,PHD,MPH, Principal Investigator — Monash University
Locations (1):
- Monash Centre for Health Research and Implementation, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Menon K, Cameron JD, de Courten M, de Courten B. Use of carnosine in the prevention of cardiometabolic risk factors in overweight and obese individuals: study protocol for a randomised, double-blind placebo-controlled trial. BMJ Open. 2021 May 13;11(5):e043680. doi: 10.1136/bmjopen-2020-043680. PMID 33986049